CLINICAL TRIAL: NCT06980064
Title: Wearable Devices Assist in the Detection, Screening, and Management of Major Diseases in Middle-aged and Elderly Populations: a Multicenter Randomized Controlled Trial
Brief Title: Wearable Devices Assist in the Detection, Screening, and Management of Major Diseases in Middle-aged and Elderly Populations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Geriatric Hospital of Nanjing Medical University (Other); The Affiliated Hospital of Yangzhou University (Unknown); Shanghai Health and Medical Center (Unknown); Weifang Hospital of Traditional Chinese Medicine (Unknown); CR & WSICO general hospital (Unknown); Xunxian People's Hospital (Unknown)
Responsible Party: Principal Investigator, Zhang Cuntai, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2024S212
Record Dates: First submitted 2025-05-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Coronary Stenosis; Cerebral Arterial Diseases; Hypertension; Parkinson Disease; Heart Failure; Peripheral Arterial Occlusive Disease; Thyroid Dysfunction
MeSH Terms: conditions — Coronary Stenosis; Cerebral Arterial Diseases; Hypertension; Parkinson Disease; Heart Failure; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (AI smartwatch assisted diagnosis) (Experimental): Participants in the intervention group will be required to wear a smartwatch continuously for 24 hours. After this period, the collected data will be processed using a pre-trained foundational model for disease diagnosis, generating preliminary diagnostic suggestions. General pratitioners will then integrate these smartwatch-derived findings with clinical interviews and aforementioned baseline examination results to formulate a final diagnosis.
  Interventions: Diagnostic Test: Smartwatch + GP
- Control group (general pratitioner only) (Active Comparator): Participants in the control group will not wear smart watches. General pratitioners will base their diagnoses solely on clinical interviews and the aforementioned baseline examinations.
  Interventions: Diagnostic Test: GP only

INTERVENTIONS:
Diagnostic Test: Smartwatch + GP — Participants in the intervention group will be required to wear a smartwatch continuously for 24 hours. After this period, the collected data will be processed using a pre-trained foundational model for disease diagnosis, generating preliminary diagnostic suggestions. GPs will then integrate these smartwatch-derived findings with clinical interviews and aforementioned baseline examination results to formulate a final diagnosis.
  Arms: Intervention group (AI smartwatch assisted diagnosis)
Diagnostic Test: GP only — GPs will make diagnosis with clinical interviews and aforementioned baseline examination results to formulate a final diagnosis.
  Arms: Control group (general pratitioner only)

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of wearable devices (Huawei smartwatches) in aiding the detection, and screening of major diseases (e.g., coronary artery disease, hypertension) in middle-aged and elderly populations aged 40-69 years with cardiovascular risk factors (e.g., smoking, diabetes, hypertension, dyslipidemia). The main questions it aims to answer are:

Does AI-assisted diagnosis using wearable device data improve the detection rate of coronary artery stenosis (CAD-RADS ≥3) compared to standard physician assessment without AI assistance?

Does the intervention reduce the incidence of coronary artery disease-related events (e.g., angina, myocardial infarction) within one year?

Researchers will compare the intervention group (AI model-assisted diagnosis based on Huawei smartwatch data) with the control group (standard assessment) to determine if the AI-aided smartwatch approach enhances diagnostic accuracy and clinical outcomes.

Participants will:

（Intervention group）Wear a Huawei smartwatch for 24 hours to collect physiological data (e.g., PPG signals, heart rate, motion).

Undergo baseline assessments, including medical history review, physical exams, and laboratory tests.

Receive a preliminary diagnosis from a general practitioner.

Complete a follow-up evaluation after one year to track cardiovascular events and other disease outcomes.

Undergo coronary CTA if suspected of coronary stenosis.

ELIGIBILITY:
The inclusion criteria are as follows:

1. Aged more than equal to 40 years, less than 69 years.
2. Having at least one of the following conditions (with one risk factor for cardiovascular and cerebrovascular diseases):

   ① Male ≥ 55 years old, female ≥ 65 years old; ② Smokers or those who quit smoking within the past 3 months prior to the visit; ③ Diabetes (type 1 or 2); ④ Hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg) or currently taking antihypertensive medication; ⑤ Dyslipidemia: total cholesterol ≥ 5.18mmol/L, triglycerides ≥ 1.70mmol/L, high-density lipoprotein<1.04mmol or low-density lipoprotein ≥ 3.37mmol/L; ⑥ hsCRP>3.0 mg/L; ⑦ 10-year ASCVD risk of 20% or more (calculated according to the formula designed in the PREVENT study)
3. Agree to receive coronary CTA if suspected to have coronary artery stenosis.
4. Voluntarily joined and signed the informed consent.

The exclusion criteria:

1. Previously diagnosed with CAD or considered moderate to severe coronary stenosis (CAD-RADS grade 3 or above: stenosis degree of 50% or above) through coronary CTA or coronary angiography examination.
2. Pregnant women or women planning to become pregnant within the next year.
3. During the onset of the disease and needs in-hospital treatment.
4. Tattoos or other substances that affect optical signals on the wrist.
5. Severe arrhythmia patients, including third degree atrioventricular block, ventricular escape rhythm, severe sinus bradycardia, sick sinus syndrome, supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, ventricular fibrillation, ventricular flutter.
6. Physical disability, blindness, and deafness.
7. Allergic history of contrast agent containing iodine.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary heart disease | From enrollment to the diagnosis, generally within 1 week
  According to the results of coronary computed tomography angiography , coronary heart disease is diagnosed if the stenosis of the coronary artery exceeds 50% (CAD-RADS grade 3 and above).

SECONDARY OUTCOMES:
Major adverse cardiovascular events | From enrollment to 1 year of follow-up
  Major adverse cardiovascular events, including myocardial infarction, stroke, aortic dissection, cardiac arrest and death from baseline to 1 year of follow-up

OTHER OUTCOMES:
Detection rate of other major chronic diseases | From enrollment to the diagnosis, generally within 1 week
  All relevant diseases will be diagnosed according to relevant guidelines, including cerebral vascular stenosis (cerebral artery computed tomography angiography), hypertension (blood pressure measurement), nocturnal hypertension (blood pressure measurement), heart failure (echocardiogram), cardiomyopathy (echocardiogram), peripheral arterial disease (vascular ultrasonography), thyroid dysfunction (thyroid function test), systemic lupus erythematosus (symptom and laboratory tests), Parkinson's disease (symptom) and sleep apnea syndrome (polysomnography).

CONTACTS AND LOCATIONS:
Overall Officials: Cuntai Zhang, PhD, Study Chair — Wuhan TongJi Hospital

IPD SHARING:
Plan to Share IPD: No
According to data policy of Huawei and Tongji hospital, individual level data will not be shared.